CLINICAL TRIAL: NCT03258970
Title: No Association Between Vitamin C and E Supplementation, Frailty, and Grip Strength Over Five Years: The CoLaus Study
Acronym: CoLaus
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Pedro Marques-Vidal, Associate professor, Centre Hospitalier Universitaire Vaudois
Other Study IDs: 2
Record Dates: First submitted 2017-08-14; First posted 2017-08-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Frail Elderly Syndrome
Keywords: vitamin supplement; Vitamin C; Vitamin E

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, blood and DNA samples available, but not used in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational cohort study — taking vitamin supplements

SUMMARY:
To assess the cross-sectional and 5-year prospective association between self-reported vitamin C+E dietary supplementation and markers of grip strength and frailty in community-dwelling Swiss adults.

DETAILED DESCRIPTION:
Participants were drawn from the Colaus study, a prospective study designed to evaluate the prevalence of cardiovascular risk factors (CVRFs) and identify genetic determinants of these risk factors in an adult Swiss population. Details of the sampling procedure have been previously published (22) and can be located online (http://www.colaus.ch).

Recruitment for the baseline Colaus study began in June 2003 and ended in May 2006, enrolling 6733 participants. The first follow-up was performed between April 2009 and September 2012, 5.5 years on average after the collection of baseline data. The information collected was similar to that in the baseline examination but included questions regarding food consumption and physical activity for the first time. The second follow-up was performed between May 2014 and July 2016, 10.7 years on average after the collection of baseline data and applied similar methods to those in the first follow-up. For this study, data from the first and the second follow-ups were used.

All participants were examined in the morning after a fast of at least 8 hours. They were surveyed about their personal and family history of cardiovascular disease, CVRFs, and cardiovascular treatment. They also specified all prescribed and nonprescribed drugs used in the last 4 weeks, including dietary and vitamin supplements.

Vitamin supplement use Vitamin supplement use and dietary intake were evaluated using a self-administered, semi-quantitative food frequency questionnaire (FFQ). This FFQ includes 3 questions regarding the intake of vitamin C, vitamin E, and multivitamins and was previously validated in the nearby Geneva population (23, 24). In short, this questionnaire computes the previous 4 weeks' dietary intake and comprises 97 distinct food items that account for more than 90% of intake of calories, proteins, fat, carbohydrates, alcohol, cholesterol, vitamin D, and retinol and 85% of fibre, carotene, and iron. There does not yet exist an FFQ in Switzerland that can assess dietary intake for an entire year (25). Thus, this FFQ provides the most accurate dietary assessment available. The FFQs were completed by participants prior to their visits so the questionnaires could be reviewed by trained investigators in person.

Vitamin C+E users were defined as those who reported consumption of at least 0.5/day of either vitamin C or vitamin E supplements on the FFQ. As there are few single-vitamin supplements available in Switzerland and many MVM can contain either vitamin C or vitamin E or both, the investigators also considered MVM for sensitivity analysis. As many participants failed to provide the exact brand name of the MVM, it was not possible to calculate the exact intake of vitamin C or vitamin E (5). Vitamin D and/or calcium supplements were coded separately and were not included in the MVM category since most vitamin D and/or calcium supplements were prescribed for management of osteoporosis in women.

Other covariates Subjects were considered smokers if they smoked at the time of the interview; former smokers were defined as smokers who had quit smoking no matter how long before their interview; never smokers were defined as those who had never smoked. Educational level was categorized as low (primary), middle (apprenticeship or high school), and high (university) for highest completed level of education. Physical activity was assessed with a self-reported questionnaire previously validated in a population living in Geneva (28). This questionnaire considers the category and duration of 70 different forms of (non)professional activities and sports from the previous 7 days. Sedentary status was defined as expending more than 90% of daily energy expenditures in activities less intense than moderate- and high-intensity (defined by expending at least 4 times one's basal metabolic rate) (29, 30).

Body weight and height were measured while participants stood without shoes in light indoor attire. Body weight was measured in kilograms to the nearest 100 g using a Seca® scale (Hamburg, Germany) that was frequently calibrated. Height was measured to the nearest 5 mm using a Seca® (Hamburg, Germany) height gauge. Body composition was examined with electrical bioelectrical impedance using the Bodystat 1500 analyzer (Isle of Man, UK) that has been previously validated (31).

Other dietary (non-vitamin) supplements were obtained from the drug questionnaire given to all participants and include substances such as shark cartilage, cod liver oil, or plant extracts not registered as phytotherapy in the Swiss drug compendium.

ELIGIBILITY:
Inclusion criteria Participation in the first follow-up of the CoLaus study Exclusion criteria for the cross-sectional study

1. missing grip strength;
2. missing covariates
3. missing or suspicious body fat values Further exclusion criteria for the prospective analysis
4. did not complete the second follow-up
5. missing grip strength at the second follow-up.

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All inhabitants of Lausanne city, Switzerland, aged 35 to 75 at the time of the Baseline study (2003-2006)
Sampling Method: Probability Sample
Enrollment: 2711 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
Grip strength | Between April 2009 and September 2012, and 5.5 years afterwards
  Grip strength was assessed using the Baseline® Hydraulic Hand Dynamometer (Fabrication Enterprises Inc, Elmsford, NY, USA) with the subject seated, shoulders adducted and neutrally rotated, elbow flexed at 90°, forearm in neutral position, and wrist between 0 and 30° of dorsiflexion per American Society of Hand Therapists's guidelines (26). Three measurements were performed successively with the subject's right hand, and the highest value (expressed in kg), along with the participant's dominant hand choice, was recorded.

SECONDARY OUTCOMES:
Low grip strength | Between April 2009 and September 2012, and 5.5 years afterwards
  Grip strength was categorized as low (defined as frail in this study) or normal according to the Fried criteria, which also considers sex and body mass index (BMI).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vollenweider, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois; Gérard Waeber, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Firmann M, Mayor V, Vidal PM, Bochud M, Pecoud A, Hayoz D, Paccaud F, Preisig M, Song KS, Yuan X, Danoff TM, Stirnadel HA, Waterworth D, Mooser V, Waeber G, Vollenweider P. The CoLaus study: a population-based study to investigate the epidemiology and genetic determinants of cardiovascular risk factors and metabolic syndrome. BMC Cardiovasc Disord. 2008 Mar 17;8:6. doi: 10.1186/1471-2261-8-6. PMID 18366642